CLINICAL TRIAL: NCT01441102
Title: A Pilot Phase I/II Study for the Evaluation of Dextromethorphan as a Microglia Inhibitor in the Treatment of Diabetic Macular Edema (MiDME2)
Brief Title: Dextromethorphan for Diabetic Macular Edema
Acronym: MiDME2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110244; 11-EI-0244 (Other: NIH CNS IRB)
Record Dates: First submitted 2011-09-24; First posted 2011-09-27 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2017-01

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; Microglia; Dextromethorphan
MeSH Terms: interventions — Dextromethorphan; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dextromethorphan hydrobromide (Experimental)
  Interventions: Drug: Dextromethorphan hydrobromide

INTERVENTIONS:
Drug: Dextromethorphan hydrobromide — Participants instructed to take 60 mg dextromethorphan capsules orally two times a day for 24 months.
  Other Names: Delsym; Creomulsion; Benylin

SUMMARY:
Background: Many people with diabetes have macular edema (swelling) at the back of the eye. Macular edema can cause loss of vision. Studies suggest that inflammation may be involved in the swelling. A drug called dextromethorphan may help prevent the inflammation and the swelling. Dextromethorphan is approved for use as a cough medicine, but it has not been studied to see if it can help in diabetic macular edema.

Objectives: To see if dextromethorphan can help treat diabetic macular edema.

Eligibility: Individuals at least 18 years of age who have diabetic macular edema in at least one eye.

Design:

* This study lasts 2 years, and will require at least 14 visits to the National Eye Institute outpatient clinic. Study visits will be every month for the first 2 months and then every other month. Each visit will take about 2 to 4 hours.
* Participants will be screened with a physical exam, medical history, eye exam, and blood tests. One eye with macular edema will be chosen as the study eye for testing.
* Participants will take dextromethorphan twice a day, about 12 hours apart, for 2 years. A study diary will help keep track of the date, time, and number of pills taken.
* Participants will have study visits once a month for the first 2 months and then every other month for the rest of the study. Each study visit will involve eye exams and blood and urine tests.
* Four months after starting the study medication, participants may have laser surgery or other treatments for the macular edema, if it is needed.

DETAILED DESCRIPTION:
Objective:

Diabetic retinopathy (DR) is one of the leading causes of blindness in the United States. A frequent manifestation of DR is diabetic macular edema (DME) for which the only proven treatment is laser photocoagulation. In the retina, microglia are capable of migrating through the retina to sites of inflammation to associate closely with neurons and the vasculature, and are key cellular players in the mediation of processes of chronic inflammation implicated in DME. For these reasons, microglia represent a promising cellular target for forms of therapy that limit the deleterious inflammatory changes found in DR. The objective of this study is to investigate the safety and efficacy of dextromethorphan as a microglia inhibitor in participants with DME.

Study Population:

Eligibility criteria include presence of diabetic retinopathy with retinal thickening due to diabetic macular edema within 3000 μm of the center of the macula as measured by optical coherence tomography (OCT), and visual acuity better than 20/200 in the study eye.

Design:

Five participants will be initially enrolled in this unmasked pilot study. However, up to an additional three participants may be enrolled to account for participants who withdraw from the study prior to receipt of six months of study treatment. Participants will take an oral dose of 60 mg of dextromethorphan twice daily for 24 months. During each visit, participants will have their visual acuity measured and will undergo OCT testing to measure retinal thickness. Beginning at the Month 4 visit, participants will be assessed for worsening disease defined as loss of ≥ 15 Early Treatment Diabetic Retinopathy Study (ETDRS) letters of vision compared to baseline or a ≥ 50% increase in total central retinal thickness as measured by OCT. Individual participants deemed to have worsening disease may stay on the study and continue to receive study medication, but will be allowed to receive focal laser therapy for any amenable leaking microaneurysms and/or anti-vascular endothelial growth factor (VEGF) intravitreal injections (such as bevacizumab or ranibizumab) at the discretion of the treating physician. Additionally, beginning at the Month 6 visit, participants will be eligible for treatment, with either focal laser or anti-VEGF injections if they have center-involving macular edema.

Outcome Measures:

The primary outcome is the change in retinal thickness measured by OCT at 6 months compared to baseline. Secondary outcomes include the change in retinal thickness as measured by OCT at 12, 18 and 24 months compared to baseline, change in best-corrected visual acuity (BCVA) at 6, 12, 18 and 24 months compared to baseline, change in mean macular sensitivity as measured by microperimetry at 6, 12, 18 and 24 months compared to baseline, as well as changes in fluid leakage in the macula as demonstrated by fluorescein angiography at 6, 12, 18 and 24 months compared to baseline. Safety outcomes include the number and severity of systemic and ocular toxicities, and adverse events.

ELIGIBILITY:
Inclusion Criteria

1. Participant is 18 years of age or older.
2. Participant must understand and sign the protocol's informed consent document.
3. Female participants of childbearing potential must not be pregnant or breast-feeding, must have a negative urine pregnancy test within 24 hours prior to initiation of study medication and must be willing to undergo urine pregnancy tests throughout the study.
4. Female participants of childbearing potential and male participants able to father children must have (or have a partner who has) had a hysterectomy or vasectomy, be completely abstinent from intercourse or must agree to practice two acceptable methods of contraception throughout the course of the study and for one week after study medication discontinuation. Acceptable methods of contraception include:

   * hormonal contraception (i.e., birth control pills, injected hormones, dermal patch or vaginal ring),
   * intrauterine device,
   * barrier methods (diaphragm, condom) with spermicide, or
   * surgical sterilization (hysterectomy or tubal ligation).
5. Participant must agree to notify the study investigator or coordinator if any of his/her doctors initiate a new medication during the course of this study.
6. Participant must agree not to take medications containing dextromethorphan during the course of this study.
7. Participant must have normal renal function and liver function, or have mild abnormalities no greater than grade 1 as defined by the Common Terminology Criteria for Adverse Events v4.0 (CTCAE).
8. Participant has a diagnosis of diabetic mellitus (type 1 or type 2). Any one of the following will be considered to be sufficient evidence that diabetes is present:

   * Current regular use of insulin for the treatment of diabetes;
   * Current regular use of oral anti-hyperglycemia agents for the treatment of diabetes;
   * Documented diabetes by American Diabetes Association (ADA) and/or World Health Organization (WHO) criteria.
9. Participant has documented hemoglobin A1C 12% or less within one month of baseline.

   * Participants with elevated hemoglobin A1C but within the 12% or less cutoff will undergo appropriate evaluation, and unstable patients will be excluded according to the investigator's best medical judgment.
   * Participant agrees to refrain from consuming grapefruit juice, grapefruits and Seville oranges at any time while s/he is enrolled in this study.
10. Participant has at least one eye that meets the study eye criteria listed below.

Exclusion Criteria

1. Participant is in another investigational study and actively receiving another study medication for diabetic macular edema (DME).
2. Participant is unable to comply with study procedures or follow-up visits.
3. Participant has a known hypersensitivity to sodium fluorescein dye.
4. Participant has a condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control).

   • Patients in poor glycemic control who, within the last four months, initiated intensive insulin treatment (a pump or multiple daily injections) or plan to do so in the next four months should not be enrolled.
5. Participant has a history of chronic renal failure requiring dialysis or kidney transplant.
6. Participant has a history of hepatitis or liver failure.
7. Participant has an allergy or hypersensitivity to dextromethorphan or levorphanol.
8. Participant is taking or has taken within the last 14 days any medication that could adversely interact with dextromethorphan such as selective serotonin reuptake inhibitors (SSRIs) or monoamine oxidase inhibitors (MAOIs) including but not limited to the following: almotriptan; amitriptyline; amoxapine; bromocriptine; buspirone; cabergoline; citalopram; clomipramine; desipramine; desvenlafaxine; dihydroergotamine; doxepin; duloxetine; eletriptan; ergoloid mesylates; ergotamine; escitalopram; fluoxetine; fluvoxamine; frovatriptan; imipramine; isocarboxazid; linezolid; lithium; maprotiline; meperidine; methylergonovine; milnacipran; mirtazapine; moclobemide; naratriptan; nefazodone; nortriptyline; paroxetine; phenelzine; procarbazine; promethazine; protriptyline; rasagiline; rizatriptan; SAMe (S-adenosylmethionine); selegiline; sertraline; sibutramine; St. Johns wort; sumatriptan; tapentadol; tramadol; tranylcypromine; trazodone; trimipramine; tryptophan; venlafaxine; vilazodone; zolmitriptan.
9. Participant has a blood pressure of > 180/110 (systolic above 180 OR diastolic above 110).

   • If blood pressure is brought below 180/110 by anti-hypertensive treatment, a patient can become eligible.
10. Participant has a history of treatment with systemic anti-vascular endothelial growth factor (VEGF) agents or steroids within three months prior to study entry.

Study Eye Inclusion Criteria

1. Best-corrected visual acuity (BCVA) Early Treatment Diabetic Retinopathy Study (ETDRS) score of 34 letters or better (i.e., 20/200 or better).
2. Definite retinal thickening due to diabetic macular edema, based on clinical examination, that is not refractory to further therapy as based on the investigator's clinical judgment.
3. Retinal thickening due to DME within 3000 μm of the center of the macula, as measured by Spectral optical coherence tomography (OCT).
4. Media clarity, pupillary dilation and patient cooperation sufficient for adequate fundus photographs.

Study Eye Exclusion Criteria

1. Macular edema is considered to be due to a cause other than diabetic macular edema.

   An eye should not be considered eligible if:
   * The macular edema is considered to be related to cataract extraction; or
   * Clinical exam and/or OCT suggest that vitreoretinal interface disease (e.g., a taut posterior hyaloid or epiretinal membrane) is the primary cause of the macular edema.
2. An ocular condition is present such that, in the opinion of the investigator, visual acuity would not improve from resolution of macular edema (e.g., foveal atrophy, pigmentary changes, dense subfoveal hard exudates, non-retinal condition).
3. An ocular condition is present (other than diabetic retinopathy (DR) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass Syndrome, etc.).
4. Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by three lines or more (i.e., cataract would be reducing acuity to 20/40 or worse if eye was otherwise normal).
5. History of panretinal scatter photocoagulation (PRP) within four months prior to study entry.
6. History of prior pars plana vitrectomy within six months prior to study entry.
7. History of major ocular surgery (including cataract extraction, scleral buckle, any intraocular surgery, etc.) within three months prior to study entry.
8. History of Yttrium aluminium garnet (YAG) capsulotomy performed within two months prior to study entry.
9. History of treatment within three months prior to enrollment with any drug that has not received regulatory approval at the time of study entry, such as intravitreal or periocular steroids or intravitreal anti-VEGF agents.

Choice of Study Eye in Cases of Bilateral Disease

If both eyes of a participant meet the criteria described above, the following will be used to determine the study eye:

1. If one eye is treatment-naïve and the other is not, the treatment-naïve eye will be chosen as the study eye.
2. If both eyes are treatment-naïve, the eye with the better visual acuity will be chosen as the study eye.
3. If both eyes are treatment-naïve and are equivalent, the choice of study eye will be determined at the investigator's discretion after consultation with the participant.
4. If both eyes have been previously treated, the choice of study eye will be determined at the investigator's discretion after consultation with the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-08; Primary Completion 2014-06 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A Cukras, MD, PhD, Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kempen JH, O'Colmain BJ, Leske MC, Haffner SM, Klein R, Moss SE, Taylor HR, Hamman RF; Eye Diseases Prevalence Research Group. The prevalence of diabetic retinopathy among adults in the United States. Arch Ophthalmol. 2004 Apr;122(4):552-63. doi: 10.1001/archopht.122.4.552. PMID 15078674
- [Background] Klein R, Klein BE, Moss SE, Davis MD, DeMets DL. The Wisconsin epidemiologic study of diabetic retinopathy. IV. Diabetic macular edema. Ophthalmology. 1984 Dec;91(12):1464-74. doi: 10.1016/s0161-6420(84)34102-1. PMID 6521986
- [Background] Ferris FL 3rd, Patz A. Macular edema: a major complication of diabetic retinopathy. Trans New Orleans Acad Ophthalmol. 1983;31:307-16. No abstract available. PMID 6623578
- [Result] Valent DJ, Wong WT, Chew EY, Cukras CA. Oral Dextromethorphan for the Treatment of Diabetic Macular Edema: Results From a Phase I/II Clinical Study. Transl Vis Sci Technol. 2018 Dec 17;7(6):24. doi: 10.1167/tvst.7.6.24. eCollection 2018 Nov. PMID 30584490
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-EI-0244.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five participant study; however, up to an additional three participants may be enrolled to account for participants who withdraw from the study prior to receipt of six months of study treatment.
Period: Overall Study
Arm/Group | Dextromethorphan Hydrobromide
Started | 7 (Two participants withdrew prior to Month 6; therefore, two additional participants were enrolled.)
Completed | 4
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 58.57 [47.00 to 66.00]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Retinal Thickness in the Study Eye at 6 Months Compared to Baseline
Description: Retinal thickness was assessed by spectral-domain optical coherence tomography (Cirrus HD-OCT; Carl Zeiss Meditec, Dublin, CA), a non-invasive imaging technique that uses long-wavelength light to capture micrometer-resolution cross-sectional images from biological tissue. The participant's eye that met the study eye eligibility criteria was selected as the study eye. For cases in which both eyes met the study eye eligibility criteria, the study eye was selected according to the "choice of study eye in cases of bilateral disease" selection criteria outlined in the eligibility criteria. The eye not chosen as the study eye is referred to as the "fellow eye."
Time Frame: Baseline and 6 months
Population: Two participants withdrew from the study prior to the 6-month visit.
Measure: Mean (Standard Deviation); unit: percentage change in retinal thickness
Units Other Than Participants: Eyes
Arm/Group | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
percentage change in retinal thickness | -7.89 (15.18)

2. Secondary Outcome: Percentage Change in Retinal Thickness in the Study Eye at 12 Months Compared to Baseline
Description: Retinal thickness was assessed by spectral-domain optical coherence tomography (Cirrus HD-OCT; Carl Zeiss Meditec, Dublin, CA), a non-invasive imaging technique that uses long-wavelength light to capture micrometer-resolution cross-sectional images from biological tissue. Changes in OCT will be calculated using the ETDRS grid. Attention will be directed to changes in retinal thickness as measured by OCT in each of the 9 subfields of the grid.
Time Frame: Baseline and 12 Months
Measure: Mean (Standard Deviation); unit: percentage change in retinal thickness
Units Other Than Participants: eyes
Arm/Group | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 4
Number analyzed (eyes) | 4
percentage change in retinal thickness | 6.54 (26.96)

3. Secondary Outcome: Percentage Change in Retinal Thickness in the Study Eye at 18 Months Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and 18 Months
Measure: Mean (Standard Deviation); unit: percentage change in retinal thickness
Units Other Than Participants: eyes
Arm/Group | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 4
Number analyzed (eyes) | 4
percentage change in retinal thickness | -0.99 (19.11)

4. Secondary Outcome: Percentage Change in Retinal Thickness in the Study Eye at 24 Months Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and 24 Months
Measure: Mean (Standard Deviation); unit: percentage change in retinal thickness
Units Other Than Participants: eyes
Arm/Group | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 4
Number analyzed (eyes) | 4
percentage change in retinal thickness | -7.44 (18.33)

5. Secondary Outcome: Change in Best-corrected Visual Acuity (BCVA) in the Study Eye at 6 Months Compared to Baseline
Description: Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters, the equivalent Snellen measurement is 20/20.
Time Frame: Baseline and 6 Months
Population: Two participants withdrew from the study prior to the 6-month visit.
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: Eyes
Arm/Group | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
ETDRS letters | 0.60 (11.44)

6. Secondary Outcome: Change in Best-corrected Visual Acuity (BCVA) in the Study Eye at 12 Months Compared to Baseline
Description: as for outcome 5
Time Frame: Baseline and 12 Months
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: Eyes
Arm/Group | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 4
Number analyzed (Eyes) | 4
ETDRS letters | 1.50 (15.02)

7. Secondary Outcome: Change in Best-corrected Visual Acuity (BCVA) in the Study Eye at 18 Months Compared to Baseline
Description: as for outcome 5
Time Frame: Baseline and 18 Months
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: Eyes
Arm/Group | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 4
Number analyzed (Eyes) | 4
ETDRS letters | 4.00 (10.74)

8. Secondary Outcome: Change in Best-corrected Visual Acuity (BCVA) in the Study Eye at 24 Months Compared to Baseline
Description: as for outcome 5
Time Frame: Baseline and 24 Months
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: Eyes
Arm/Group | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 4
Number analyzed (Eyes) | 4
ETDRS letters | 5.50 (12.58)

9. Secondary Outcome: Number of Study Eyes Demonstrating a Decrease in the Area of Late Leakage, as Measured by Fluorescein Angiography (FA), at 6 Months Compared to Baseline
Description: Fluorescein angiography (FA) images were obtained via a standard digital imaging system (OIS, Sacramento, CA) at baseline and at Month 6, Month 12, Month 18, and Month 24. Three retinal specialists independently graded the area of late fluorescein leakage (at approximately 10 minutes) using a region-of-interest tool in an image analysis software package (NIH ImageJ, Bethesda, MD).
Time Frame: Baseline and 6 Months
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 5
Number analyzed (eyes) | 5
eyes | 4

10. Secondary Outcome: Number of Study Eyes Demonstrating a Decrease in the Area of Late Leakage, as Measured by Fluorescein Angiography (FA), at 12 Months Compared to Baseline
Description: as for outcome 9
Time Frame: Baseline and 12 Months
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 4
Number analyzed (eyes) | 4
eyes | 3

11. Secondary Outcome: Number of Study Eyes Demonstrating a Decrease in the Area of Late Leakage, as Measured by Fluorescein Angiography (FA), at 18 Months Compared to Baseline
Description: as for outcome 9
Time Frame: Baseline and 18 Months
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 4
Number analyzed (eyes) | 4
eyes | 2

12. Secondary Outcome: Number of Study Eyes Demonstrating a Decrease in the Area of Late Leakage, as Measured by Fluorescein Angiography (FA), at 24 Months Compared to Baseline
Description: as for outcome 9
Time Frame: Baseline and 24 Months
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 4
Number analyzed (eyes) | 4
eyes | 4

13. Secondary Outcome: Changes in Mean Macular Sensitivity in the Study Eye at 6 Months Compared to Baseline
Description: Microperimetry was used to assess macular sensitivity.
Time Frame: Baseline and 6 Months
Measure: Mean (Standard Deviation); unit: dB
Units Other Than Participants: eyes
Arm/Group | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 5
Number analyzed (eyes) | 5
dB | -2.1 (3.10)

14. Secondary Outcome: Changes in Mean Macular Sensitivity in the Study Eye at 12 Months Compared to Baseline
Description: Microperimetry was used to assess macular sensitivity.
Time Frame: Baseline and 12 Months
Measure: Mean (Standard Deviation); unit: dB
Units Other Than Participants: eyes
Arm/Group | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 4
Number analyzed (eyes) | 4
dB | -3.7 (3.44)

15. Secondary Outcome: Changes in Mean Macular Sensitivity in the Study Eye at 18 Months Compared to Baseline
Description: Microperimetry was used to assess macular sensitivity.
Time Frame: Baseline and 18 Months
Measure: Mean (Standard Deviation); unit: dB
Units Other Than Participants: eyes
Arm/Group | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 4
Number analyzed (eyes) | 4
dB | -4.9 (3.97)

16. Secondary Outcome: Changes in Mean Macular Sensitivity in the Study Eye at 24 Months Compared to Baseline
Description: Microperimetry was used to assess macular sensitivity.
Time Frame: Baseline and 24 Months
Measure: Mean (Standard Deviation); unit: dB
Units Other Than Participants: eyes
Arm/Group | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 2
Number analyzed (eyes) | 2
dB | -3.9 (3.54)

17. Secondary Outcome: Number of Participants Withdrawn From the Study Therapy Due to Vision Loss or Adverse Events
Time Frame: Duration of the study, up to 24 months
Measure: Number; unit: participants
Arm/Group | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 7
participants | 1

ADVERSE EVENTS:
Time Frame: Duration of the study, up to 24 months per participant
Arm/Group | Dextromethorphan Hydrobromide
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dextromethorphan Hydrobromide (N=7)
Vitreous haemorrhage (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dextromethorphan Hydrobromide (N=7)
Vitreous haemorrhage (Eye disorders) | 2 (2)
Malaise (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Furuncle (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Feeling jittery (General disorders) | 1 (1)
Renal function test abnormal (Investigations) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Episcleritis (Eye disorders) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Arthropod Bite (Injury, poisoning and procedural complications) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Iridocyclitis (Eye disorders) | 1 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Eye Pain (Eye disorders) | 1 (1) — Event reported as pain in the right eye.
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Vitreous floaters (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes